CLINICAL TRIAL: NCT03848988
Title: A Descriptive Analysis of Back Pain Patient's Seeking Care at Chiropractic Academic Teaching Clinics Using the STarT Back Screening Tool: Cross-sectional Survey and Chart Review
Brief Title: Descriptive Analysis: STarT Back Screening Tool: Cross-sectional Survey & Chart Review
Acronym: STarT Back
Status: Completed | Type: Observational
Sponsor: Parker University (Other)
Collaborators: Baylor Scott and White Health (Other); Private Practitioner (Unknown)
Responsible Party: Sponsor
Other Study IDs: Parker19_001
Record Dates: First submitted 2019-02-18; First posted 2019-02-21 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Back Pain
Keywords: Chiropractic; Screening tool; Teaching
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Keele STarT Back SCreening Tool (KSB) is a practical and validated bio-psychosocial questionnaire that stratifies lower back pain patients into 3 risk groups (low, medium, high), with suggested treatment guidelines for each grouping. The 9-question KSB has been used in chiropractic practice to help guide medical decision making, but its use in chiropractic teaching environments has been limited.

DETAILED DESCRIPTION:
All new LBP patients between the ages of 18-65 years presenting to a chiropractic teaching clinic in Dallas, TX between March 05, 2018 and April 06, 2018 were asked to complete the KSB questionnaire. No introduction of the KSB was given to students or faculty. For all patients that completed the KSB, a chart review of the first 4 weeks of care was completed to retrieve patient follow-up information and treatment provided, including: self-reported LBP on a 10-point numerical rating scale (NRS), region of spinal manipulation therapy (SMT), and active rehabilitation provided.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age of 18-65 years old.

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Accepted all genders, biological and/ or self-preference.
Study Population: New LBP patients presenting to a chiropractic teaching clinic in Dallas, TX
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-04-06 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
Chiropractic care Questionnaire | 4 weeks
  Nine question Keele STarT Back questionnaire to identify treatment options for individuals with low, moderate, and high risk low back pain. A 10 point numerical rating scale (NRS) was used to with 0-4 being low risk, 5 being moderate risk, and 6-10 being high risk.

SECONDARY OUTCOMES:
Low back pain self reported | 4 weeks
  Oswestry low back pain scale/ tool: 10 point scale with 0 being no pain and 10 being excruciating pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Parker University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided